CLINICAL TRIAL: NCT01648153
Title: A Single Blind (Sponsor-unblinded), Placebo-controlled, Parallel-group Study to Investigate the Efficacy and Safety of GSK1070806 in the Treatment of Obese Subjects With T2DM.
Brief Title: Investigate the Efficacy and Safety of GSK1070806 in Obese Subjects With T2DM
Acronym: T2DM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 116378
Record Dates: First submitted 2012-07-12; First posted 2012-07-24 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus
Keywords: Efficacy; Obese; T2DM; IL-18; Monoclonal antibody (mAb)
MeSH Terms: conditions — Diabetes Mellitus; Obesity | interventions — GSK1070806; Sodium Chloride

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- GSK1070806 0.25mg/kg (Active Comparator): TwoIV administrations of 0.25mg/kg GSK1070806 4weeks apart
  Interventions: Biological: GSK1070806
- GSK1070806 5mg/kg (Active Comparator): Two IV administrations of 5mg/kg of GSK1070806 4 weeks apart
  Interventions: Biological: GSK1070806
- Placebo (Saline) (Placebo Comparator): Two IV administrations of saline 4 weeks apart
  Interventions: Other: Placebo (saline)

INTERVENTIONS:
Biological: GSK1070806 — To investigate the efficacy and biomarker changes of GSK1070806 after 0.25mg/kg IV administration
  Arms: GSK1070806 0.25mg/kg
Other: Placebo (saline) — To compare the efficacy and biomarker changes between placebo and active groups
  Arms: Placebo (Saline)
Biological: GSK1070806 — To investigate the efficacy and biomarker changes of GSK1070806 after 5mg/kg IV administration
  Arms: GSK1070806 5mg/kg

SUMMARY:
GSK1070806 is a humanised IgG1/kappa antibody which is directed against the soluble cytokine interleukin-18 (IL-18). The aims of this placebo controlled study are to evaluate the efficacy, safety, tolerability, pharmacokinetics and pharmacodynamics of GSK1070806 in obese subjects with Type 2 diabetes mellitus (T2DM), and to gain a better understanding of the mechanism by which GSK1070806 exerts its therapeutic effects.

DETAILED DESCRIPTION:
The study will be a randomised, single-blind (sponsor-unblinded), placebo-controlled, study to investigate the efficacy, safety, tolerability, pharmacokinetics and pharmacodynamics of repeat intravenous infusions (2 doses 4-weeks apart) of GSK1070806 in obese patients with T2DM. The primary objective of the study will be to assess improvements in fasting and postprandial glucose control. This will be a parallel-group study in 30 obese subjects with T2DM who are poorly controlled on metformin monotherapy (HbA1C>7% but <9.5%), and who have levels of microalbuminuria indicative of progressive kidney disease i.e. 30-300mg/L albumin in urine or ACR ≥3.5 mg/mmol (female) or ≥2.5 mg/mmol (male) and ≤30mg/mmol. There will be three treatment groups comprising two active and one placebo arm with 10 subjects per dose group. The study contains a broad range of biomarker assessments, the purpose of which is to evaluate the mechanistic basis by which GSK1070806 exerts its therapeutic benefit in subjects with T2DM.

Subjects will be randomised into one of the three treatment groups where they will receive two intravenous infusions of GSK1070806 or placebo twenty-eight days apart. A MMT challenge will be conducted on Day 1, Day 29, Day 57 and Day 85 for evaluation of the primary endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of T2DM as determined by a responsible physician based on a medical evaluation including medical history, physical examination, and laboratory tests, with onset at least 6 months prior to Screening.
2. Male or female between 18 and 70 years of age inclusive, at the time of signing the informed consent.
3. HbA1c levels ≥ 7.0 % and ≤ 9.5%; at Screening.
4. On a stable dose of monotherapy with metformin for three months prior to screening, and at a total daily dose greater than or equal to 1000 mg for at least 2 months prior to dosing.
5. Fasting plasma glucose level < 13.3 mmol/L (240 mg/dL) at screening.
6. Obese with BMI ≥ 30 kg/m2, and < 40 kg/m2.
7. Presence of microalbuminuria: 30-300mg/L albumin in urine or Albumin Creatinine Ratio (ACR) ≥ 3.5 mg/mmol (female) or ≥2.5 mg/mmol (male) and ≤ 30 mg/mmol (female and male)..
8. The subject is capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
9. A female subject is eligible to participate if she is of:

   * Non-childbearing potential
   * Child-bearing potential and agrees to use an acceptable form of contraception.
10. Male subjects must agree to use one of the contraception methods listed
11. ALT < 2xULN; alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
12. Single or Average QTc, QTcB or QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.

Exclusion Criteria:

1. Current evidence, or history within the last 7 days, of an influenza-like illness as defined by fever (>38°C) and two or more of the following symptoms: cough, sore throat, runny nose, sneezing, limb / joint pain, headache, vomiting / diarrhoea in the absence of a known cause, other than influenza.
2. Use of anti-inflammatory drugs including corticosteroids, chronic maintenance therapy with NSAIDs, anti-Tumor Necrosis Factor (anti-TNF) or anti-Interleukin-1 (anti-IL1) within 60 days prior to dosing.
3. Current evidence of ongoing or acute infection, history of repeated, chronic or opportunistic infections (e.g. recurrent folliculitis, other cutaneous infections or repeated pneumonia) or history of a serious bacterial infection within 6 months of randomisation.
4. History of malignancy or significant cardiac, pulmonary, metabolic, renal, hepatic, or gastrointestinal conditions.
5. History chronic granulomatous infections, such as of Mycobacterium tuberculosis or any other previous Mycobacterium infection.
6. Creatinine clearance less than 60ml/min
7. Screens positive of Hepatitis B surface antigen, Hepatitis C antibody or Human Immunodeficiency Virus (HIV)
8. History of a severe allergic reaction, anaphylaxis or immunodeficiency.
9. Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
10. A positive pre-study drug/alcohol screen.
11. History of regular alcohol consumption within 6 months of the study
12. The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
13. Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
14. Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication.
15. History of sensitivity to any of the study medications, or components thereof
16. Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
17. Pregnant females as determined by positive serum or urine hCG test at screening.
18. Lactating females.
19. Unwillingness or inability to follow the procedures outlined in the protocol.
20. Subject is mentally or legally incapacitated.
21. Subject has received a live attenuated vaccine(s) within 30 days of randomisation or will require vaccination with a live attenuated vaccine prior to the end of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-08; Primary Completion 2013-09 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in fasting plasma glucose and weighted mean glucose AUC (0-4hrs) post-Mixed Meal Test (MMT) | Up to 85 days after the first does
  To evaluate the efficacy of two repeat intravenous dose administrations of GSK1070806 in subjects with T2DM

SECONDARY OUTCOMES:
Safety and tolerability parameters include: adverse events, clinical laboratory tests, electrocardiograms (ECGs), and vital signs | Up to 210 days after the first dose
  To evaluate the safety and tolerability of two repeat intravenous dose administrations of GSK1070806 in obese subjects with T2DM
Change from baseline in % HbA1c, fasting blood insulin, and C-peptide levels; change from baseline in weighted mean insulin, and C-peptide levels [AUC (0-4hrs)] post-MMT and derived measures of insulin sensitive | Up to 85 days after the first dose
  To evaluate the effect of two repeat intravenous dose administrations of GSK1070806 on additional markers of efficacy, in obese subjects with T2DM
AUC(0-τ) | Up to 210 days after the first dose
  To evaluate the plasma PK of repeat intravenous doses of GSK1070806 in obese subjects with T2DM
Serum levels of free IL-18 and drug bound IL 18 | Up to 210 days after the first dose
  To investigate the effect of repeat intravenous doses of GSK1070806 on free and drug bound IL 18 levels (if measurable) in obese subjects with T2DM.
Change from baseline in serum and/or plasma levels of biomarkers of inflammation (e.g. hs-CRP, and IL-6) and metabolic disease (e.g. adiponectin, fructosamine, total cholesterol, high-density lipoprotein (HDL)/low-density lipoprotein (LDL), triglycerides | Up to 85 days after the first dose
  To explore the pharmacodynamic (PD) effect of repeat intravenous doses of GSK1070806 on biomarkers of inflammation and metabolic disease
Change from baseline in waist circumference and BMI | Up to 85 days after the first dose
  To investigate the effect of repeat intravenous doses of GSK1070806 on body composition in obese subjects with T2DM
Cmax | Up to 210 days after the first dose
  To evaluate the plasma PK of repeat intravenous doses of GSK1070806 in obese subjects with T2DM
Tmax | Up to 210 days after the first dose
  To evaluate the plasma PK of repeat intravenous doses of GSK1070806 in obese subjects with T2DM
after the second dose λz | Up to 210 days after the first dose
  To evaluate the plasma PK of repeat intravenous doses of GSK1070806 in obese subjects with T2DM
t1/2 | Up to 210 days after the first dose
  To evaluate the plasma PK of repeat intravenous doses of GSK1070806 in obese subjects with T2DM

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- Spain (9):
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Alzira/Valencia
  - GSK Investigational Site, Granada
  - GSK Investigational Site, La Roca Del Valles (Barcelona)
  - GSK Investigational Site, Lleida
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Petrer, Alicante
  - GSK Investigational Site, Santander
- United Kingdom (3):
  - GSK Investigational Site, Birmingham, Warwickshire
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, Dundee

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] McKie EA, Reid JL, Mistry PC, DeWall SL, Abberley L, Ambery PD, Gil-Extremera B. A Study to Investigate the Efficacy and Safety of an Anti-Interleukin-18 Monoclonal Antibody in the Treatment of Type 2 Diabetes Mellitus. PLoS One. 2016 Mar 1;11(3):e0150018. doi: 10.1371/journal.pone.0150018. eCollection 2016. PMID 26930607
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 116378 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116378 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116378 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116378 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116378 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116378 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116378 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register